CLINICAL TRIAL: NCT03649204
Title: Effect of a Hybrid Rehabilitation Program on Walking, Quality of Life and Cardiovascular Risk in People With Peripheral Arterial Disease (HY-PAD): A Pilot Randomized Controlled Trial
Brief Title: Effect of a Hybrid Rehabilitation Program on Walking, Quality of Life & Cardiovascular Risk in People With PAD
Acronym: HY-PAD
Status: Recruiting | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: AFP Innovation Fund (Other)
Responsible Party: Sponsor
Other Study IDs: 774
Record Dates: First submitted 2018-08-23; First posted 2018-08-28 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: HY-PAD — Hybrid intervention that includes supervised on-site and home-based components in people with PAD

SUMMARY:
Peripheral arterial disease (PAD), a disabling condition, affects 800,000 Canadians. People with PAD suffer from poor quality of life due to leg pain, which makes walking difficult. They also have a high risk of heart disease. In November of 2017, the University of Ottawa Heart Institute (UOHI) launched Canada's first specific walking rehabilitation and cardiovascular risk reduction program dedicated to patients with PAD.

An on-site, supervised exercise program to improve walking endurance and quality of life in PAD has been shown to be successful. However many patients are not able to participate in the on-site program due to barriers such as transportation, parking, or other commitments. Recently, a home-based walking program has also been shown to significantly improve walking endurance and quality of life among people with PAD. It was decided that a hybrid program, that has a short on-site program followed by a home-based program may allow more patients to participate and have the highest chance of success.

The goal is to develop a new hybrid program for medical care in PAD patients in order to: (a) improve their walking distance, (b) improve their quality of life and (c) improve their cardiovascular risk.

As part of this study the investigators will enrol 25 participants with PAD. Participants will be studied at baseline (before their first on-site class) and at 3 month follow up (after their last home program phone call).

ELIGIBILITY:
Inclusion Criteria:

* Intermittent claudication with PAD documented by:

  * ABI ≤0.90 or >1.40;(14) or
  * Anatomic evidence of lower extremity arterial stenosis ≥50% (by lower extremity angiography, CT angiography, MR angiography or ultrasound)
* Ability to participate in the study (ability to walk)
* Willingness to provide informed consent

Exclusion Criteria:

* They have had previous lower extremity amputation
* They are unable to walk
* They have critical limb ischemia or open lower extremity wounds.
* Patient is unable to read and understand English or French
* Patient is unable, in the opinion of the qualified investigator or referring physician, to comprehend and participate in the exercise intervention.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who enroll in the UOHI PAD walking program
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-07-09 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
6MWT | at 3 month follow up
  Improvements (increase) in 6 minute walk test total walking distance (meters) after 3 months

SECONDARY OUTCOMES:
Improvements in quality of life | at 3 month follow up
  Improvement (increase) in accelerometer-measurement MVPA (meters/week), and Improvements in total claudicant distance (meters)
improvements in Walking Impairment Questionnaire | at 3 month follow up
  Increase in WIQ (Walking Impairment Questionnaire) scores Responses are ranked on a scale of 0 to 4, (0=unable to do, 4=no difficulty)

CONTACTS AND LOCATIONS:
Overall Officials: Thais Coutinho, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada